CLINICAL TRIAL: NCT06526572
Title: Measuring Pain Perception in Patients With Symptomatic Acute Pulpitis and Resistant to Inferior Alveolar Nerve Block Using NRS and Brain Waves
Brief Title: Pain Measured by NRS and EEG in Acute Pulpitis
Status: Recruiting | Type: Observational
Sponsor: Cleveland Dental Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CDIENDO0007
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Acute Pulpitis
Keywords: Acute pulpits; Electroencephalography; Numerical rate scale; Inferior Alveolar Nerve Block
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- symptomatic acute pulpitis: Patients with symptomatic acute pulpitis who are resistant to inferior alveolar nerve block (IANB)
  Interventions: Diagnostic Test: Brain wave analysis using electroencephalography (EEG).; Diagnostic Test: Numerical rate Scale (NRS)

INTERVENTIONS:
Diagnostic Test: Brain wave analysis using electroencephalography (EEG). — Asessment of pain with objective neurophysiological assessment through brain wave analysis using electroencephalography (EEG).
Diagnostic Test: Numerical rate Scale (NRS) — Asessment of pain with the subjective numercal rate scale method (NRS

SUMMARY:
The aim of the proposed study is to investigate and comprehensively understand pain perception in patients diagnosed with symptomatic acute pulpitis who are resistant to inferior alveolar nerve block (IANB).

The study aims to achieve this by utilizing a dual approach that combines subjective self-reporting of pain intensity using the Numeric Rating Scale (NRS) with objective neurophysiological assessment through brain wave analysis using electroencephalography (EEG).

By integrating these two methods, the study seeks to explore potential correlations between self-reported pain scores and neural responses recorded through EEG, providing insights into the pain experience of this specific patient population.

Ultimately, the goal of the study is to enhance the understanding of pain perception mechanisms in individuals with symptomatic acute pulpitis resistant to IANB and potentially guide the development of more effective and personalized pain management strategies for these patients.

ELIGIBILITY:
Inclusion Criteria:

Adults aged [18-50 years]. Clinically diagnosed with symptomatic acute pulpitis based on dental examination and radiographic findings.

Demonstrates resistance to inferior alveolar nerve block (IANB). Willing and able to provide informed consent to participate in the study. Able to communicate effectively in the language used for study procedures.

Exclusion Criteria:

Individuals with known neurological or psychiatric disorders affecting pain perception.

Pregnant individuals or those breastfeeding at the time of the study. History of severe allergies or adverse reactions to local anesthetics or EEG gel.

Presence of significant medical conditions that may contraindicate dental procedures or EEG recordings.

Individuals taking medications that could significantly affect pain perception (e.g., strong analgesics, sedatives).

Any contraindications for dental procedures or EEG recordings as determined by the study's dental and medical professionals.

Inability to understand and follow study instructions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults male or females aged [18-50 years], Clinically diagnosed with symptomatic acute pulpitis based on dental examination and radiographic findings. They are medically free. They are willing and able to provide informed consent to participate in the study. They are able to communicate effectively in the language used for study procedures.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | 3 months
  Changes in alpha brain waves in patients with acute pulpitis and resistant to alveolar nerve block injection
Numerical Rate Scale (NRS) | 3 months
  Measuring pain perception using NRS (Scale 0-10 where 0 is no pain and 10 is the most unbearable pain) in patients with acute pulpitis and resistant to alveolar nerve block injection.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A hashem, PhD, Study Director — CDI Centro Diagnostico Italiano S.p.A
Locations (1):
- Cleveland Dental Institute, Cleveland, Ohio, United States